CLINICAL TRIAL: NCT04327245
Title: Effect of Intake of Stevia and D-tagatose Sweeteners on Glycemia, Peptide C and Appetite-satiety in Women With Insulin Resistance
Brief Title: To Compare the Effects of Non-nutritive Sweeteners Intake in Woman With Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Sociedad Chilena de Diabetes y Endocrinología (SOCHED) (Unknown)
Responsible Party: Principal Investigator, Verónica Sambra Vásquez, Co-Director, University of Chile
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: SOCHED
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Insulin Resistance; Hyperinsulinism
Keywords: High-Intensity Sweeteners; Non-Nutritive Sweeteners; Stevia rebaudiana; C-Peptide; Blood Glucose
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism | interventions — tagatose

STUDY DESIGN:
Intervention Model Description: The experimental design was developed 3 times. Each intervention was performed separately for a minimum period of 7 days out and a maximum of 14 days, depending on the availability of the experimental subjects. Cross treatment design (crossover) each women serves as its own control The first intervention corresponded to the control group, in order to maintain the ignorance of the type of sweetener they were receiving, between day 7 or maximum 14 days post-intervention the order of the test of the NNS was reversed. Therefore, during the second or third intervention they were given to drink water with D-tagatose or stevia respectively
Who Masked: Participant
Masking Description: the participant has no knowledge of the intervention assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention ingest a 5000 mg of D-tagatose (Experimental): Intervention: Women with resistance insulin who ingest a 5000 mg of D-tagatose. D-tagatose is a sweetener of natural origin, low in calories (1.5 kcal / g) and with a sweetness power of 0.9.e.
  Interventions: Other: Intervention ingest a 5000 mg of D-tagatose
- No Intervention: Intervention ingest a water (control group) (No Intervention): Woman with resistance insulin who ingest a water (control group)
- Intervention ingest a 15,3 mg of stevia (Experimental): Intervention: Woman with resistance insulin who ingest a 15,3 mg of stevia (steviol glycosides). The word "stevia" refers to the whole plant of Stevia rebaudiana Bertoni (SRB), only some of the components of the stevia leaf are sweet.
  Interventions: Other: Intervention ingest a 15,3 mg of stevia

INTERVENTIONS:
Other: Intervention ingest a 5000 mg of D-tagatose — Woman with resistance insulin who ingest a 5000 mg of D-tagatose. D-tagatose is a sweetener of natural origin, low in calories (1.5 kcal / g) and with a sweetness power of 0.9.
  About 20 to 25% of the ingested D-tagatose is absorbed and metabolized in the liver, the rest is fermented by the microbiota producing short chain fatty acids.
  Arms: Intervention ingest a 5000 mg of D-tagatose
Other: Intervention ingest a 15,3 mg of stevia — Woman with resistance insulin who ingest a 15,3 mg of stevia (steviol glycosides). The word "stevia" refers to the whole plant of Stevia rebaudiana Bertoni (SRB), only some of the components of the stevia leaf are sweet. Steviol glycosides are up to 300 times sweeter than sucrose, do not provide calories and can be used as a substitute for sucrose or as a non-nutritive sweetener alternative. Your allowable daily intake is 4 mg / kg / body weight (expressed as steviol)
  Arms: Intervention ingest a 15,3 mg of stevia

SUMMARY:
ABSTRACT

Introduction: There is no current data about the effects of non-nutritive sweeteners (NNS) about important factors, such as the energy intake, appetite and its relationship in people with insulin resistance when tasting sweet. It is highly relevant to compare the effects of NNS intake, such as, stevia (steviol glycosides) and D-tagatose, previous to a 75-gram oral glucose tolerance test (OGTT) on glycaemic and C-peptide responses in women with insulin resistance.

Objective: To compare the effects of non-nutritive sweeteners intake: stevia (steviol glyco-sides) and sucralose previous to OGTT on appetite, glycemia and C-peptide plasmatic concentrations in women with insulin resistance.

Methods: Thirty-three women with T2DM were studied in 3 different moments and they received 3 treatments: pre-load of water or D-tagatose or stevia and then offered to consume a 75-gram oral glucose tolerance test. Blood samples were obtained to measure the dependent variables, glycemic at times -10, 0, 30, 60, 90, 120 and 180 minutes and C-peptide at times -10, 30, 90, 120 and 180 minutes. The analogue visual scale questionnaires (VAS) was conducted every 30 minutes in order to obtain the results of the depend variables: appetite and wish of specific type of food in a subjective way; appetite, satiety, relax, wish to eat any food, craving for something sweet, craving for something salty, something tasty, something fatty. Through food provided ad libi-tum (objective appetite), were obtained the results of: energy, carbohydrates, proteins and lipid intakes. The statistical analysis applied included the Shapiro-Wilk's Normality test, repeated measures ANOVA to assess differences among treatments, Friedman's test followed by Wilcoxon test corrected by Bonferroni as needed. The degree of association between variables was conducted using the Pearson's or Spearman's correlation coefficient tests, as requested. A probability value p <0.05 was considered significant.

DETAILED DESCRIPTION:
Protocol The experimental design was developed 3 times. Each intervention was performed separately for a minimum period of 7 days out and a maximum of 14 days, depending on the availability of the experimental subjects. Cross treatment design (crossover) each women serves as its own control The first intervention corresponded to the control group, in order to maintain the ignorance of the type of sweetener they were receiving, between day 7 or maximum 14 days post-intervention the order of the test of the NNS was reversed. Therefore, during the second or third intervention they were given to drink water with D-tagatose or stevia respectively. For each intervention a check list was followed.

Subjects were asked to maintain their normal diet between study days and abstain from strenuous exercise and alcohol intake for 24 hours before each evaluation. The subjects attended with an 8-hour fast, without having ingested medication, to the sampling room of the Pharmacy Faculty, University of Valparaís. The study was only begun if they had a capillary glycemia <100%, measured through a glucometer.

Then, they were asked to answer the analogue visual scale (VAS) questionnaire and an intravenous catheter was installed in the antecubital vein to take the blood samples at "time -10". Immediately, they were given to drink 60 ml of water or 60 ml of water with 5000 mg of D-tagatose or an equivalent volume with 15,3 mg of stevia (steviol glycosides), which they had to consume in less than 2 minutes.

After 10 minutes, at "time 0" immediately after the second blood sample, the individuals consumed a 75-gram oral glucose tolerance test (OGTT).

The following blood samples were taken at times 30, 60, 90, 120 and 180 minutes after "time 0". In total, 28 ml of blood was extracted, in each time the glycemia and C-peptide were determined (4 ml was taken at a time).

In addition, VAS questionnaires were applied every 30 minutes, from "time -10" to 180 minutes for appetite determinations.

After completing the extraction of blood samples at 180 minutes and removing the intravenous catheter, the subjects were offered a meal for 30 minutes, which consisted of a variety of foods of high acceptability, previously weighed and fractionated.

Statistic analysis The normal distribution of the variables was determined by the Shapiro-Wilk test. The natural logarithm was applied to the parameters without normal distribution. The variables were expressed as mean ± standard deviation or median plus interquartile interval (Q1-Q3). The statistical significance between the differences in plasma glucose concentrations, area under the curve (AUC) of glycaemia, energy intake and macronutrients by treatment (preload water, D-tagatose and stevia), was evaluated through Anova of repeated samples . To analyze the differences between plasma concentrations and AUC of C-peptide and glycaemia per treatment (preload water, D-tagatose and stevia), Friedman's test was used, followed by Wilcoxon and adjusted by Bonferroni.

To identify the relationships between glycemic responses and intake of food at will (energy intake and macronutrients by treatment, preload water, D-tagatose and stevia), the Pearson correlation factor was used, in contrast to C-peptide response and the visual analogue scale (VAS) and food intake at will per treatment Spearman's correlation factor was used.

The statistical analysis was performed with the SPSS 20.0 computer program (SPSS Inc., Chicago Illinois). A p <0.05 was considered statistically significant for all the analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Woman with Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) ≥ 2,5
* Body Mass Index (BMI) between 18.5 to 34.9 kg / m2
* Stable doses of oral contraceptive
* cigarette smoking <5 units / day
* Women on metformin treatment were allowed with the requirement of discontinuation for a period of four weeks prior to study initiation.

Exclusion Criteria:

* sex male
* pregnant or lactating women
* women with diseases, conditions or medications that provoke hyperinsulinism or that alter the glucidic metabolism, the postprandial hormonal response, appetite and / or satiety
* those who carry out moderate to intense physical activity three or more times a week for more than 30 minutes at a time
* those with the use of vitamin supplements or antioxidants
* Women with an allergy or aversion to the sweeteners used in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
glycemic response in blood | Three hours
  Area under the curve was built for each subjects after steviol or D-tagatose or water intake.

SECONDARY OUTCOMES:
C-peptide response in blood | Three Hours
  Area under the curve was built for each subjects after steviol or D-tagatose or water intake.

OTHER OUTCOMES:
The analogue visual scale questionnaires (VAS) | 30 minutes
  Used to measure the appetite sensation includes three characteristic concepts; hunger, fullness and satiety. Understanding hunger for: vital and indispensable physiological need to nourish our body; Fullness: State that invites to stop eating; and satiety as: Sensation of satisfaction. The visual analog scale (VAS) of 10 cm in length will be used with words anchored at each end, which expresses the most positive rating (value 10 cm) and the most negative (0 cm). It will be used to evaluate hunger, satiety, fullness, prospective food consumption, desire to eat something sweet, salty, tasty or fatty, scale whose reference is "Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord 2000; 24 (1): 38-48 was conducted every 30 minutes in order to obtain the results of the depend variables.
Through food provided ad libitum (objective appetite) | 30 minutes
  were obtained the results of: energy, carbohydrates, proteins and lipid intakes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sambra V, Vicuna IA, Priken KM, Luna SL, Allendes DA, Godoy PM, Novik V, Vega CA. Acute responses of stevia and d-tagatose intake on metabolic parameters and appetite/satiety in insulin resistance. Clin Nutr ESPEN. 2022 Jun;49:217-224. doi: 10.1016/j.clnesp.2022.04.018. Epub 2022 Apr 22. PMID 35623816